CLINICAL TRIAL: NCT00543907
Title: Outcomes of a Deep Inferior Epigastric Perforator Flap Program
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Bernard T. Lee, Professor of Surgery, Beth Israel Deaconess Medical Center
Other Study IDs: 2007P000232
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; DIEP flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre programmatic development: Patients who have undergone mastectomy for breast cancer prior to implementation of the deep inferior epigastric perforator flap microsurgical breast reconstruction program
- Post programmatic development: Patients who have undergone mastectomy for breast cancer after implementation of the deep inferior epigastric perforator flap microsurgical breast reconstruction program

SUMMARY:
The purpose of this study is to analyze an institution's experience with starting a subspecialized DIEP flap program.

DETAILED DESCRIPTION:
The purpose of this study is to analyze an institution's experience with starting a subspecialized DIEP flap program and to determine whether other hospitals would benefit from instituting a similar program. Prior studies have compared the outcome from a DIEP flap program with that of TRAM flaps within the same center. Other studies have calculated the cost of a DIEP flap and its complication rate. However, no one has examined the overall effects of a subspecialized reconstruction program and its impact on a health center. In this study, we will determine if the institutionalization of a DIEP flap program has increased our center's rate of breast reconstruction, as well as evaluate its outcomes and overall financial viability.

ELIGIBILITY:
Inclusion Criteria:

* Intraductal carcinoma
* Lobular carcinoma
* Infiltrating ductal carcinoma
* Paget's disease
* BRCA positive

Exclusion Criteria:

* Inflammatory carcinoma of the breast

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who have undergone mastectomy for breast cancer between 1999 and 2008 at the BIDMC.
Sampling Method: Non-Probability Sample
Enrollment: 977 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
complication rate | 6 years
  complication rate

SECONDARY OUTCOMES:
reconstruction rate | 6 years
  reconstruction rate
patient satisfaction | 6 years
  Breast Q, Michigan Breast Outcomes Survey

CONTACTS AND LOCATIONS:
Overall Officials: Bernard T Lee, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No